CLINICAL TRIAL: NCT06173349
Title: A Phase I Microtrial With PLZ4-Coated Paclitaxel-Loaded Micelles (PPM) in Patients With Recurrent or Refractory Non-Myoinvasive Bladder Cancer
Brief Title: PLZ4-Coated Paclitaxel-Loaded Micelles for the Treatment of Patients With Recurrent or Refractory Non-Muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mamta Parikh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Mamta Parikh, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#309; NCI-2023-10047 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UCDCC#309 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Non-Muscle Invasive Bladder Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PLZ4-coated paclitaxel loaded micelles (PPM) (Experimental): Patients receive PPM intravesically over 1 hour QW for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, or PET, and cystoscopy with biopsy at screening and follow up and undergo collection of blood samples throughout the trial.
  Interventions: Drug: PLZ4-coated paclitaxel loaded micelles (PPM)

INTERVENTIONS:
Drug: PLZ4-coated paclitaxel loaded micelles (PPM) — Given PLZ4-coated paclitaxel loaded micelles intravesically
  Other Names: Paclitaxel; PPM

SUMMARY:
This phase I trial tests the safety, tolerability and effectiveness of PLZ4-coated paclitacel-loaded micelles (PPM) in treating patients with non-muscle invasive bladder cancer that has come back after a period of improvement (recurrent) or that does not respond to treatment (refractory). PPM is a bladder cancer-specific nanoparticle that can specifically target and deliver treatment to the tumor cells in the bladder. PPM contains paclitaxel, which is a drug that kills tumor cells or keeps them from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the safety and tolerability of PPM administered through intravesical instillation.

SECONDARY OBJECTIVES:

I. Evaluate tumor response at 6 weeks after completion of PPM intravesical therapy.

II. Assess event-free survival rate at 12 months.

OUTLINE:

Patients receive PPM intravesically over 1 hour once a week (QW) for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET), and cystoscopy with biopsy at screening and follow up and undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up at 3 weeks, 6 weeks, and then every 3 months per standard of care for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non muscle invasive bladder cancer (NMIBC), defined as noninvasive papillary carcinoma (Ta), carcinoma in situ (CIS) or carcinoma invading the subepithelial connective tissue (T1), determined via transurethral resection of bladder tumor (TURBT) within 3 months of enrollment
* Participant must have Bacillus Calmette Guerin (BCG)-unresponsive NMIBC or intolerance of treatment with BCG. BCG-unresponsive disease is defined as being at least one of the following:

  * Persistent or recurrent CIS alone or with recurrent Ta/T1 (noninvasive papillary disease/tumor invades the subepithelial connective tissue) disease within 12 months of completion of adequate BCG therapy
  * Recurrent high-grade Ta/T1 disease within 12 months of completion of adequate BCG therapy
  * T1 high-grade disease at the first evaluation following an induction BCG course. In this context, adequate BCG therapy is defined as at least one of the following:

    * At least five of six doses of an initial induction course plus at least two of three doses of maintenance therapy
    * At least five of six doses of an initial induction course plus at least two of six doses of a second induction course
* Refuse or intolerant of a radical cystectomy recommended by the treating urologist as the standard next therapy per American Urological Association (AUA) guideline
* Age ≥ 18 years at time of consent
* Performance status: Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Patient with life expectancy greater than 24 months
* No concurrent radiotherapy, chemotherapy, or other immunotherapy for bladder cancer. No BCG or other intravesical treatment within 4 weeks
* No scheduled radiotherapy, chemotherapy, other immunotherapy, or surgery before the scheduled response evaluation
* Recovery from prior treatment side effects that might interfere with the study treatment, in the judgment of the investigator
* Absolute neutrophil count (absolute granulocyte count [AGC]/absolute neutrophil count [ANC]) ≥ 1,500/µL
* Platelets ≥ 100,000/µL (Patients may be transfused to meet this requirement)
* Hemoglobin ≥ 8 g/dL (Patients may be transfused to meet this requirement)
* Calculated glomerular filtration rate (GFR) ≥ 30 mL/min
* Total bilirubin ≤ 2.0 × institutional upper limit of normal (ULN) (< 3 × ULN for patients with Gilbert's syndrome)
* Aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP) ≤ 3.0 × institutional ULN
* Adequate pulmonary function by clinical assessment with no clinical signs of severe pulmonary dysfunction
* Participants of childbearing potential must agree to using adequate contraception (e.g., hormonal or barrier method of birth control; abstinence, an intrauterine device) for the duration of study participation (including dosing interruptions) and up to 3 months after last study treatment; or be surgically sterilized (e.g., hysterectomy, tubal ligation, or vasectomy)
* Ability to understand and willingness to sign an informed consent form
* Ability and willingness to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Existence of cancer at the upper urinary tract
* Concurrent use of other investigational agents
* Evidence of regional and/or distant metastasis
* NYHA (New York Heart Association) class III or IV heart failure, uncontrollable supraventricular arrhythmias, any history of a ventricular arrhythmia, or other clinical signs of severe cardiac dysfunction
* Symptomatic congestive heart failure (CHF), severe/unstable angina pectoris, or myocardial infarction within 6 months prior to study entry
* Patient has an intractable bleeding disorder (e.g., coagulation factors deficiencies, Von Willebrand Disease)
* Patient taking medications that affect coagulation, such as aspirin (though, aspirin 81 mg oral once daily is allowed), Coumadin/Warfarin, heparin, low molecular weight heparin, direct thrombin inhibitors, and direct factor Xa inhibitors. Other nonsteroidal antiinflammatory drugs (NSAIDs) are allowed as long as they are discontinued the day before therapy
* History or evidence of uncontrollable central nervous system (CNS) disease
* Active systemic infection requiring parenteral antibiotic therapy
* Women who are pregnant or breast feeding
* Any other malignancy diagnosed within 3 years of trial entry with the exception of the following:

  * Basal or squamous cell skin cancers, or
  * Noninvasive cancer of the cervix, or
  * Any other cancer deemed to be of low-risk for progression or patient morbidity during trial period, such as localized prostate cancer after definitive treatment and prostate-specific antigen (PSA) less than 0.2 ng/mL
* Any condition that would prohibit the understanding or rendering of informed consent
* Any condition that in the opinion of the investigator would interfere with the participant's safety or compliance while on trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | From first dose of study medication through 12 months after the last dose
  Number of participants experiencing treatment-related AEs, classified by severity and graded according to the NCI CTCAE v5.0

SECONDARY OUTCOMES:
Tumor response | At 6 weeks after the last dose of study medication
  Assessment of response will be based on visual evaluation (cystoscopy), biopsy of remaining lesion (where technically feasible) and urine cytology.
Event-free survival | From first dose of study medication to first documentation of objective tumor progression, disease recurrence, bladder resection or irradiation, other anti-bladder cancer therapy, or to death due to disease progression, assessed at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Parikh, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States